CLINICAL TRIAL: NCT01837199
Title: Clinical and Microbiological Effects of Adjunctive Metronidazole Plus Amoxicillin in the Treatment of Generalized Chronic Periodontitis: Smokers Versus Non-Smokers.
Brief Title: MTZ Plus AMX in the Treatment of Smokers and Non-smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Marcelo Faveri, DDS, PhD., University of Guarulhos
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SISNEP/726
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Periodontitis; Smoking
Keywords: Periodontal disease; Scaling and root planing; Metronidazole; Amoxicillin; Generalized chronic periodontitis; Periodontal treatment
MeSH Terms: conditions — Chronic Periodontitis; Smoking; Periodontal Diseases | interventions — Metronidazole; Amoxicillin; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoking (Experimental): Metronidazole plus Amoxicillin
  Interventions: Drug: Metronidazole plus Amoxicillin
- Non-Smoking (Experimental): Metronidazole plus Amoxicillin
  Interventions: Drug: Metronidazole plus Amoxicillin

INTERVENTIONS:
Drug: Metronidazole plus Amoxicillin — All subjects will receive scaling and root planing combined with systemic metronidazole (400 mg) and amoxicillin (500 mg). Both antibiotics were administered T.I.D. for 14 days.
  Other Names: Metronidazole; Amoxicillin; Scaling and root planing

SUMMARY:
Randomized controlled clinical trials have demonstrated that the use of amoxicillin (AMX) and metronidazole (MTZ) as adjuncts to mechanical therapy improves the clinical and microbiological outcomes of scaling and root planing (SRP) in non-smokers and smokers with ChP. However, the effects of this antibiotic protocol have not been directly compared in non-smokers and smokers. Therefore, the aim of this study will be to compare the clinical and microbiological effects of the adjunctive use of MTZ+AMX to SRP in smokers and non-smokers subjects with chronic periodontitis (ChP). It was hypothesized that non-smokers would benefit better from this combination of therapies than the smokers.

DETAILED DESCRIPTION:
Sample size calculation:

This study is designed to compare the clinical and microbiological effects of the treatment of smoker and non-smoker subjects with SRP+MTZ+AMX. The ideal sample size to assure adequate power for this clinical trial was calculated considering differences of at least 1mm between groups for clinical attachment level (CAL) in initially deep periodontal sites (PD ≥ 7 mm). It was also determined that the standard deviation of CAL change at deep sites would be 1.0 mm based on our earlier studies of smokers and non-smokers receiving SRP combined with MTZ+AMX. Based on these calculations, it was defined that 26 subjects per group would be necessary to provide an 85% power with an α of 0.01. Considering an attrition of about 20%, it was established that at least 32 subjects should be included in each treatment group.

Experimental design and treatment protocol:

In this cohort clinical trial, subjects will be assigned according to their smoking status, into smoker and non-smoker groups. All subjects will receive SRP combined with systemic MTZ (400 mg) and AMX (500 mg). Both antibiotics will be administered T.I.D. for 14 days. Before the study begins, all subjects will receive full-mouth supragingival scaling and instruction on proper home-care techniques. They will receive the same dentifrice to use during the study period (Colgate Total). All subjects will receive full-mouth SRP performed under local anesthesia in four to six appointments lasting approximately 1h each. Treatment of the entire oral cavity will be done in 14 days. SRP will be performed by one trained periodontist using manual instruments. The antibiotic therapies will start immediately after the first session of mechanical instrumentation. The University Pharmacy will prepare the antibiotic pills and send them to the study coordinator, who will mark the code number of each subject on a set of two packs and give them to the examiner. All subjects will receive clinical and microbiological monitoring at baseline and at 3, 6 and 12 months post-therapy.

Clinical monitoring:

One calibrated examiner will perform clinical monitoring and the treatment will carried out by another clinician. Thus, the examiner and the clinician will be masked as to the nature of the treatment groups. Visible plaque (presence or absence), gingival bleeding (presence or absence), bleeding on probing (BOP; presence or absence), suppuration (presence or absence), PD (mm) and clinical attachment level (CAL, mm) will be measured at six sites per tooth (mesiobuccal, buccal, distobuccal, distolingual, lingual and mesiolingual) in all teeth, excluding third molars. The PD and CAL measurements will be recorded to the nearest millimeter using a North Carolina periodontal probe.

Microbiological Monitoring:

Subgingival plaque samples will be collected at baseline and at 3, 6 and 12 months post-SRP from nine non-contiguous interproximal sites per subject. The select sites will be randomized in different quadrants and subset according to baseline PD, three samples in each of the following categories: shallow (PD<3 mm), intermediate (PD 4-6 mm) and deep (PD>7 mm). After the clinical parameters have been recorded, the supragingival plaque will be removed and the subgingival samples will be taken with individual sterile curettes (Gracey #11-12) and immediately placed in separate Eppendorf tubes containing 0.15 ml of buffer (TE). One hundred microliters of 0.5 M sodium hydroxide (NaOH) will be added to each tube and the samples will be dispersed using a vortex mixer. The samples will be analyzed by Checkerboard DNA-DNA hybridization.

ELIGIBILITY:
Inclusion Criteria:

* Chronic periodontitis (AAP 1999);
* ≥35 years of age;
* Presence of at least 15 teeth;
* Minimum of 6 teeth with at least one site each with PD and clinical attachment level (CAL) ≥5 mm;
* At least 30% of the sites with PD and CAL ≥4 mm and bleeding on probing (BOP).
* Smokers: had smoked at least 10 cigarettes per day for a minimum of 5 years;
* Non-smokers: had never smoked.

Exclusion Criteria:

* Previous subgingival periodontal therapy;
* Pregnancy;
* Nursing;
* Systemic diseases that could affect the progression of periodontal disease (e.g. diabetes, osteoporosis);
* Long-term administration of anti - inflammatory medications;
* Need for antibiotic pre-medication for routine dental therapy;
* Continuous use of mouthrinses containing antimicrobials;
* Antibiotic therapy in the previous 6 months
* Allergy to MTZ or AMX.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean clinical attachment level change post- scaling and root planing in sites with initial probing depth ≥ 7 mm | At 3, 6 and 12 months post-therapy.

SECONDARY OUTCOMES:
Number of subjects with low, moderate and high risk for disease progression. | At 3, 6 and 12 months post-therapy
Mean full-mouth clinical attachment level. | Baseline and at 3, 6 and 12 months post-therapy
Mean full-mouth probing depth. | Baseline and at 3, 6 and 12 months post-therapy.
Mean clinical attachment level change post-scaling and root planing in sites with initial probing depth between 4-6 mm | At 3, 6 and 12 months post-therapy
Mean probing depth reduction post-scaling and root planing in sites with initial probing depth between 4-6 mm | At 3, 6 and 12 months post-therapy.
Mean probing depth reduction post-scaling and root planing in sites with initial probing depth ≥ 7 mm | At 3, 6 and 12 months post-therapy.
Mean changes in levels of the 40 bacterial species evaluated by Checherboard DNA-DNA hybridization | At 3, 6 and 12 months post-therapy.
Mean changes in proportions of the 40 bacterial species evaluated by Checherboard DNA-DNA hybridization | At 3, 6 and 12 months post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Faveri, DDS, PhD., Principal Investigator — University of Guarulhos; Magda Feres, DDS, PhD., Principal Investigator — University of Guarulhos; Luciene C Figueiredo, DDS, PhD., Principal Investigator — University of Guarulhos
Locations (1):
- University of Guarulhos, Guarulhos, São Paulo/ SP, Brazil